CLINICAL TRIAL: NCT00526357
Title: The Effect of Dietary Supplementation With Encapsulated Fish Oil on Mannitol-induced Airway Sensitivity and Inflammation in Persons With Asthma
Brief Title: Effect of Dietary Supplements With Fish Oil on Mannitol-induced Airway Sensitivity & Inflammation in Persons With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Firestone Institute for Respiratory Health (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Michael Quinn, Manager, Firestone Institute for Respiratory Health
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: R.P. #06-2750; Health Canada File No. 120532
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Asthma
Keywords: omega-3 fatty acids; asthma; airway hyperresponsiveness; inflammation
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity; Inflammation | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): Of the 24 asthmatic subjects, 12 will be enrolled who are taking beta2 agonists alone to treat their asthma
  Interventions: Drug: omega-3 fatty acid
- B (Other): Of the 24 asthmatic subjects, 12 will be enrolled who are taking beta2 agonists and inhaled steroids to treat their asthma
  Interventions: Drug: omega-3 fatty acid

INTERVENTIONS:
Drug: omega-3 fatty acid — Pharmaceutical grade fish oil administered daily in the form of 10 capsules (5 capsules b.i.d.) each containing 400mg of eicosapentaenoic acid (EPA) and 200mg docosahexanoic acid (DHA) which will equate to a daily dose of 4000 mg of EPA and 2000 mg or DHA. The matched placebo containing a 50/50 mix of soybean and corn oil will be supplied by the same manufacturer (Ocean Nutrition, Canada)
  Other Names: Meg-3, Product No. 4020EE

SUMMARY:
We wish to investigate the effects of 3 weeks of orally administered fish oil supplements on the airway sensitivity (provoking dose to cause a 15% fall in FEV1, PD15) to inhaled mannitol (AridolTM). Mannitol, an osmotic stimulus has been demonstrated as a useful model for exercise-induced asthma. We also wish to investigate if there is any associated improvement associated with selected markers of airway inflammation that can be measured in the sputum, blood, urine and exhaled breath condensate. Oral fish oil supplements have recently been demonstrated to be effective inhibitors of exercise-induced asthma, in association with an inhibition of markers of inflammation, over a 3 week treatment period. This finding has important implications in the treatment of asthma as this is a faster and more effective improvement than what is seen with inhaled corticosteroids on exercise-induced asthma. This observation requires validation and further investigation. We wish to study this in two patient groups; (a) steroid naïve asthmatics taking beta2 agonist when required and (b) asthmatics taking regular inhaled corticosteroids < 1000 mcg/day.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disorder of the airways characterized by recurrent episodes of dyspnea, wheeze and chest tightness and is associated with variable airway obstruction. Exercise-induced bronchoconstriction (EIB) is a feature specific to asthma. Exercise testing protocols have been developed to identify the presence of asthma as well as to assess asthma therapy. Airway narrowing following exercise in persons with asthma is thought to result from dry air hyperpnoea-induced dehydration of the airway surface, leading to the release of mediators from inflammatory cells residing in the airway. Regular treatment with inhaled corticosteroids inhibits the airway response to exercise by decreasing the number of inflammatory cells and thus the source of bronchoconstricting mediators. Therefore, a decrease in the source of mediator may be the reason for this eventual inhibition of the airway response to exercise.

It has recently been demonstrated that fish oil supplementation in capsule form, taken daily over three weeks, provides significant protection against EIB. This protection appears to be of equal or greater efficacy than inhaled corticosteroids treatment over a similar period. This may have positive implications in the treatment of asthma as inhaled corticosteroids are known to have some unwanted side effects. Fish oil supplementation in the high doses given in previous studies have not demonstrated any side effects and may lead to an alternative treatment, or a decrease in the dose of inhaled steroids required in the treatment of asthma.

A new bronchial provocation test using inhaled mannitol, derived from the mechanism of EIB, has been recently developed and is now registered in Australia and the European Union. Mannitol causes airway narrowing in a similar manner to exercise in persons with asthma and is effective in identifying responsiveness to inhaled corticosteroids. We wish to use inhaled mannitol as a model for EIB in an effort to further investigate the use of fish oil supplementation in the treatment of asthma. Our hypothesis is that daily orally administered encapsulated fish oil will attenuate the airway response to mannitol over a 3-week treatment period. We also wish to measure associated markers of inflammation in the blood, urine, sputum and exhaled condensate as well as monitor clinical outcomes such as symptoms and daily beta2 agonist use.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (medically or surgically postmenopausal or practicing an accepted form of barrier or hormonal contraception) subjects age 18-55.
* Stable, mild atopic asthma with forced expiratory volume in one second (FEV1) greater than 70% of predicted for age and height, and not requiring any medical treatment other than short acting inhaled beta2-agonists as required or for those on steroids, taking < 1000 mcg of inhaled corticosteroid per day.
* No recent or significant history of cigarette smoking (no smoking within six months prior to entry into the study; less than 10 pack-years cumulative history of cigarette smoking).
* Signed written informed consent to participate in the study; ability to return to the clinic for repeated visits.
* No history of asthma exacerbations or acute intercurrent respiratory illness (viral respiratory syndrome, bronchitis, pneumonia) for a four week period preceding entry into the screening phase of the study.
* Subjects who take inhales steroids regularly must demonstrate reproducibility to inhaled mannitol (PD15<1.0 doubling doses) during a 2 week run-in period.
* A PD15 to the mannitol challenge < 315mg

Exclusion Criteria:

* Significant gastrointestinal (including hepatic), hematological, cardiovascular, cerebrovascular, metabolic such as including type II diabetes or other body system disorder.
* Regular consumption of fish consisting more than 1 meal of fish per week or regular fish oil supplements during the trial and for at least 2 weeks prior to the first study visit.
* Subjects who have taken oral corticosteroids or a leukotriene receptor antagonist in 4 weeks prior to entry into the study.
* Psychosis, alcoholism, active substance abuse, or any personality disorder, which would make compliance with this protocol problematic.
* Pregnant or nursing females.
* Any other medical or social condition which, in the opinion of the investigator, could confound the interpretation of the data derived from this study.
* Subjects taking >1000 mcg of inhaled steroids daily in those subjects taking inhaled steroids.
* Subjects requiring regular anti-histamines for allergies.
* Subjects who have allergy to fish or any other ingredient in the study products.
* Subjects using anti-coagulants (warfarin, heparin)
* Subjects who have surgery planned over the course of the trial.
* Subjects who use medications to lower LDL cholesterol levels
* Subjects using non-steroidal anti-inflammatory medications (e.g., aspirin, ibuprofen)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The cumulative dose of mannitol to cause a 15% reduction in FEV1 (PD15). | 3 weeks

SECONDARY OUTCOMES:
Change following treatment in resting levels of eicosanoid metabolites in blood, urine & exhaled breath condensate (EBC). Sputum counts of eosinophils and metachromatic cells and LTB4, IL-a and TNF-a in sputum supernatant. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul M O'Byrne, MD, Principal Investigator — Firestone Institute for Respiratory Health
Locations (1):
- Firestone Institute for Respiratory Health, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Brannan JD, Bood J, Alkhabaz A, Balgoma D, Otis J, Delin I, Dahlen B, Wheelock CE, Nair P, Dahlen SE, O'Byrne PM. The effect of omega-3 fatty acids on bronchial hyperresponsiveness, sputum eosinophilia, and mast cell mediators in asthma. Chest. 2015 Feb;147(2):397-405. doi: 10.1378/chest.14-1214. PMID 25321659